CLINICAL TRIAL: NCT03299309
Title: The PRiME Study: PEP-CMV in Recurrent MEdulloblastoma/Malignant Glioma
Brief Title: PEP-CMV in Recurrent MEdulloblastoma/Malignant Glioma
Acronym: PRiME
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Landi (Other)
Collaborators: Pediatric Brain Tumor Foundation (Unknown); Annias Immunotherapeutics, Inc. (Other)
Responsible Party: Sponsor-Investigator, Daniel Landi, Assistant Professor of Pediatrics and Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00079843
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Medulloblastoma; Recurrent Brain Tumor, Childhood; Malignant Glioma
Keywords: Glioma; Medulloblastoma; PRiME; Pro00079843; Thompson; Pediatric; Landi
MeSH Terms: conditions — Medulloblastoma; Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEP-CMV (Experimental): Cytomegalovirus (CMV)-specific peptide vaccine (PEP-CMV)
  Interventions: Drug: PEP-CMV

INTERVENTIONS:
Drug: PEP-CMV — Patients receive temozolomide (TMZ) 200 mg/m2/day x 5 days. On day 20, patients will receive a Tetanus-diphtheria pre-conditioning vaccination with Td (tetanus, diphtheria toxoid, adsorbed). Immunotherapy begins the following day, on day 21, with injection of the PEP-CMV vaccine as follows: PEP-CMV Component A mixed with Montanide ISA-51 intradermally administered half in the RIGHT groin and half in the LEFT groin.
  Other Names: PEP-CMV vaccine

SUMMARY:
The primary goal of this prospective clinical trial is to evaluate the safety of PEP-CMV in patients with recurrent medulloblastoma and malignant glioma. Patients with histologically-proven medulloblastoma or malignant glioma who had received prior therapy for their initial diagnosis and subsequently had tumor recurrence/progression may be enrolled any time after recurrence/progression regardless of prior adjuvant therapy. PEP-CMV is a vaccine comprised of Component A, a synthetic long peptide (SLP) of 26 amino acid residues from human pp65. In May 2021, enrollment on the study was temporarily suspended due to delays in vialing the PEP-CMV study vaccine.

DETAILED DESCRIPTION:
Once a patient has enrolled onto this study, prior therapy will be terminated and patients will receive temozolomide 200 mg/m2/day x 5 days. If they are receiving bevacizumab at the time of enrollment, they will continue bevacizumab 10 mg/Kg every 14 days.

Patients who are ≥ 18 years of age will receive a tetanus (Td) booster at the time of enrollment. Immunotherapy begins with a Tetanus (Td) pre-conditioning vaccine delivered intradermally (i.d.) in the right groin at the site of the vaccine injection 6-24 hours prior to the first vaccine on day 21. The PEP-CMV vaccine will be administered as follows: PEP-CMV Component A mixed with Montanide ISA-51 (1:1 volume ratio) intradermally administered half in the RIGHT groin and half in the LEFT groin.

The first 3 PEP-CMV vaccines will occur every 2 weeks, then PEP-CMV vaccines will continue monthly (+/- 2 weeks) for no more than 10 years. Blood will be obtained for immune system monitoring.

In May 2021, enrollment on the study was temporarily suspended due to delays in vialing the PEP-CMV study vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 3 - 35 years old
2. Histopathologically proven previous diagnosis of medulloblastoma or Grade III or IV glioma.
3. Radiology evidence of recurrent medulloblastoma (reMB) or recurrent Grade III and IV glioma. Patients will be considered for a biopsy or resection of the recurrent/progressive tumor at the discretion of the treating neurosurgeon and neuro-oncologist.
4. Brain MRI within one month prior to enrollment.
5. Received prior therapy for their initial diagnosis prior to recurrence/progression or who are unable to receive radiation therapy due to genetic disorders that put them at significant risk for radiation-induced secondary malignancies (i.e. Gorlin's syndrome or NF1 mutation).
6. Patients with neurological deficits should have deficits that are stable for a minimum of 2 weeks prior to registration.
7. Karnofsky Performance Status (KPS) of ≥ 60% (KPS for > 10 years of age) or Lansky performance Score (LPS) of ≥ 60 (LPS for ≤ 10 years of age) assessed within 2 weeks prior to registration. Patients who are unable to walk because of paralysis but who are up in a wheel chair will be considered ambulatory for the purposes of the performance score.
8. Bone Marrow:

   * ANC (Absolute neutrophil count) ≥ 1000/µl (unsupported)*.
   * Platelets ≥ 100,000/µl (unsupported)*.
   * Hemoglobin > 8 g/dL (may be supported).
9. Renal:

   • Serum creatinine ≤ upper limit of institutional normal.
10. Hepatic:

    * Bilirubin ≤ 1.5 times upper limit of normal for age.
    * SGPT (ALT) ≤ 3 times institutional upper limit of normal for age.
    * SGOT (AST) ≤ 3 times institutional upper limit of normal for age.
11. Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
12. Signed informed consent according to institutional guidelines must be obtained prior to registration.
13. Any prior chemoradiotherapy is allowed.

Exclusion Criteria:

1. Pregnant or need to breast feed during the study period (Negative serum pregnancy test required).
2. Active infection requiring treatment or an unexplained febrile (> 101.5 degrees F) illness.
3. Known immunosuppressive disease or human immunodeficiency virus infection.
4. Patients with active renal, cardiac (congestive cardiac failure, myocardial infarction, myocarditis), or pulmonary disease.
5. Patients receiving concomitant immunosuppressive agents for medical condition.
6. Patients who need definitive radiotherapy for treatment of recurrent MB or recurrent Grade III or IV glioma.
7. Patients receiving any other investigational drug therapy.
8. Patients on corticosteroids > 0.1 mg/Kg/day (i.e. > the maximum dose of 4 mg/day).
9. Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction).
10. Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with unacceptable toxicity | 2 weeks after the 3rd PEP-CMV vaccine on the last enrolled patient
  Evaluate the safety of PEP-CMV in pediatric patients with recurrent MB or recurrent Grade III/IV glioma

SECONDARY OUTCOMES:
Mean or median change from baseline at each follow-up assessment in ELISPOT (IFN-γ) | 24 months
  Quantitate the immune response to the components of the PEP-CMV vaccine by ELISPOT
Mean or median change from baseline at each follow-up assessment in ELISA (gB-KLH) | 24 months
  Quantitate the immune response to the components of the PEP-CMV vaccine by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Landi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/